CLINICAL TRIAL: NCT00473473
Title: A Multicenter, Randomized, Double Blind, Placebo Controlled Trial to Investigate the Efficacy and Safety of the Homeopathic Remedy Kalium Bichromicum (Potassium Dichromate) to Decrease Viscosity and Amount of Sputum as Well as Time to Extubation, in Intubated Mechanically Ventilated ICU Patients.
Brief Title: Effect of the Homeopathic Remedy Kalium Bichromicum (Potassium Dichromate) on Viscosity and Amount of Sputum and Time to Extubation in Mechanically Ventilated ICU Patients.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Collaborators: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Menachem Oberbaum, Director, Center for Integrative Complementary Medicine, Shaare Zedek Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KaliBic.ICU.07
Record Dates: First submitted 2007-05-14; First posted 2007-05-15 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Mechanical Ventilation
Keywords: homeopathy; Traumeel; mechanical ventilation; secretions
MeSH Terms: interventions — Potassium Dichromate; Homeopathy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): potassium bichromate
  Interventions: Drug: Potassium Dichromate (Homeopathy)
- 2 (Placebo Comparator): placebo
  Interventions: Drug: Placebo homeopathic remedy

INTERVENTIONS:
Drug: Potassium Dichromate (Homeopathy) — twice daily with an interval of 12 hours, for a period of up to 14 days
  Arms: 1
Drug: Placebo homeopathic remedy — identical to treatment without active component
  Arms: 2

SUMMARY:
ICU-Protocol.Summary Profuse and tenacious tracheal secretions are a significant factor impeding the weaning process in mechanically ventilated patients in the intensive care unit (ICU). In homeopathy, high dilutions of plant extracts, minerals, and other biological substances are used as remedies for the treatment of illness, which is based on the "Law of Similars" (the higher the dilution, the stronger the effect). Kali Bichromicum (potassium dichromate) is a drug that is commonly used in homeopathy, mostly for conditions involving profuse, stringy, tenacious mucous and tracheal secretions. A recent randomized, double-blind, placebo-controlled study found a statistically significant effect of this remedy on improving the amount of tracheal secretion, timing to extubation and discharge from the ICU among critically ill patients, with no side effects observed.

The proposed study will compare the efficacy of Kali bichromicum 10-60 (C30) versus placebo in reducing the amount of tracheal secretions in patients intubated with a conventional endotracheal tube or tracheostomy and receiving controlled mechanical ventilation in the ICU setting. The quantity of the secretions will be studied, as well as sputum neutrophil count (using direct microscopy). Time to extubation and the need for re-intubation will also be evaluated. 56 patients over the age of 18 years treated with mechanical ventilation for at least 3 days will be recruited from the ICU departments of 4 medical centers in Israel. The preparations will be administered in the form of small pellet-like globules, which will be placed on the mucosa of the mouth, to the side of the endotracheal tube. Patients will be randomly allocated to either verum (n=28) or placebo (n=28) treatment, with the remedies administered twice daily with an interval of 12 hours, for a period of up to 14 days or until the patient is extubated. Any adverse event will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* endotracheally intubated or tracheostomy ICU patient on mechanical ventilation support for at least 3 days prior to study enrollment, who is due for Spontaneous Breathing Trial (SBT).
* profuse tenacious, stringy tracheal secretions (from 2+ to 4+)

Exclusion Criteria:

* Unstable septic patients
* Concomitant disease of the larynx and trachea obstructing the airway or inhibiting the extubation process.
* active heart disease.
* Need for catecholamines.
* Pregnancy.
* underlying neuromuscular disorder or any other condition preventing patient cooperation with voluntary coughing and expectoration of secretions.
* underlying conditions requiring continuous therapy with bronchorrheic medications (i.e. myasthenia gravis)
* Patients on home ventilation or BIPAP support
* Failure of the patient or legal guardian to give written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2008-07; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
the amount of tracheal secretions in patients intubated with a conventional endotracheal tube and receiving controlled mechanical ventilation with a respirator two days after the initiation of the study. | 14 days

SECONDARY OUTCOMES:
grade 3 tracheal secretions, number of suctionings and sputum neutrophil count on day 2; tracheal secretions on day 14/extubation; time to extubation and need for re-intubation; time to discharge; safety of of Kali bichromicums after 14 days/extubation. | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Menachem Oberbaum, M.D., Principal Investigator — Shaare Zedek Medical Center, Jerusalem, Israel; Moshe Hersch, M.D., Study Director — Intensive Care Unit, Shaare Zedek Medical Center, Jerusalem, Israel
Locations (2):
- Israel (2):
  - Intensive Care Unit, Shaare Zedek Medical Center, Jerusalem
  - Dept. of Internal Medicine, Intensive Care Unit G8, Hadassah University Hospital, Ein Kerem, Jerusalem

REFERENCES:
- [Background] Frass M, Dielacher C, Linkesch M, Endler C, Muchitsch I, Schuster E, Kaye A. Influence of potassium dichromate on tracheal secretions in critically ill patients. Chest. 2005 Mar;127(3):936-41. doi: 10.1378/chest.127.3.936. PMID 15764779